NCT04963062 Protocol 2021-0695 Version date: 8/30/2021

## Randomized Clinical Trial Evaluating the Efficiency and Safety of Holmium Laser with Moses Technology versus SuperPulsed Laser System with Thulium Laser on Renal and Ureteral Stones

Principal Investigator: Stephen Nakada, MD

University of Wisconsin-Madison, School of Medicine and Public Health, Department of Urology

NCT04963062 Protocol 2021-0695 Version date: 8/30/2021

## **Data Analysis Plan**

Statistical analyses include using appropriate categorical/continuous and parametric/non-parametric statistical test. Patient demographics (such age, gender, race ethnicity) and stone characteristics (such as stone volume, location, density) will be summarized as appropriate as continuous variables (mean and standard deviation) or categorical variables (frequency, percentage). To compare the two groups, procedural time, laser time, ablation speed, ablation efficiency, total energy used, are analyzed using Wilcoxon test. The score of quality of life survey and laser evaluation survey are analyzed using MANOVA. Complication rate is analyzed using chi-square. Statistical significance is set as two-tailed p value < 0.05 and data are analyzed using SPSS 25.